CLINICAL TRIAL: NCT02732067
Title: Death Rate in Anesthesia: a Prospective Study of Two Years Period From a Tertiary Hospital
Brief Title: Death Rate in Anesthesia, a Study in a Tertiary Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Subhi M. Alghanem, Professor of Anesthesia and Intensive Care, University of Jordan
Other Study IDs: 270/14a/tk
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Sudden Death
Keywords: Anesthesia
MeSH Terms: conditions — Death, Sudden

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: anesthesia related deaths — number of anesthetized patients who died in the perioperative period inside the hospital

SUMMARY:
Death rate in anesthesia is one of the most valuable methods to assess the safety of anesthesia practice among different types of patients.

In this study, the investigators will follow the death among patients who underwent surgery under anesthesia whether regional or general over the next two years from 2016 to 2018.

DETAILED DESCRIPTION:
Death rate in anesthesia is one of the most valuable methods to assess the safety of anesthesia practice among different types of patients. Most of the studies of death rate in anesthesia are retrospective with many drawbacks and pitfalls like absence of information in the records of the patients.

In this study, the investigators will follow the death among patients who underwent surgery under anesthesia whether regional or general over the next two years from 2016 to 2018, by examining the patients records from the hospital database and recording the events that occur to the dead patients.

The end point of this study will be anesthesia death rate inside the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent anesthesia and surgery.
* Patients who died inside the hospital.

Exclusion Criteria:

* Patient who underwent anesthesia and surgery and do not died and discharged home.
* Patients who died outside the hospital.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent anesthesia and surgery and died inside the hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
number of anesthetized patients who died in the perioperative period inside the hospital | 30 days post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Subhi M Alghanem, FFARCS, Study Chair — Jordan University
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Watters DA, Hollands MJ, Gruen RL, Maoate K, Perndt H, McDougall RJ, Morriss WW, Tangi V, Casey KM, McQueen KA. Perioperative mortality rate (POMR): a global indicator of access to safe surgery and anaesthesia. World J Surg. 2015 Apr;39(4):856-64. doi: 10.1007/s00268-014-2638-4. PMID 24841805